CLINICAL TRIAL: NCT02130310
Title: A Phase-3 Prospective, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Efficacy of CureXcell® as an Adjunct to Good Ulcer Care Measures in Treating Chronic Venous Leg Ulcers
Brief Title: Evaluation of CureXcell® in Treating Chronic Venous Leg Ulcers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Macrocure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MC-105
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Venous Leg Ulcers
Keywords: Chronic ulcers; Venous ulcers
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CureXcell® (Experimental): CureXcell® injection will be administered about every 4 weeks for up to 3 treatments, or until ulcer closure, whichever occurs first.
  Interventions: Biological: CureXcell®
- Placebo injection (Placebo Comparator): The placebo will be administered by injecting normal saline at each centimeter of the ulcer bed.
  Interventions: Other: Placebo injection

INTERVENTIONS:
Biological: CureXcell® — CureXcell® is a cell based therapy obtained from donated whole blood. The blood is collected from healthy young adults, the white blood cells are separated and then activated by hypo-osmotic shock.
  Arms: CureXcell®
Other: Placebo injection — Normal saline injected at each centimeter of ulcer bed
  Arms: Placebo injection

SUMMARY:
The primary objective is to evaluate the clinical benefit of CureXcell® as adjunct to Standard of Care in the treatment of Chronic Venous Leg Ulcers. CureXcell® is a cell based therapy, containing activated homologous white blood cells prepared from donated healthy whole blood. A total of 252 patients will be randomized to receive either CureXcell® or Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Ankle Brachial Pressure Index (ABI) ≥ 0.80
* Venous insufficiency confirmed by duplex Doppler ultrasound
* Presence of a venous leg ulcer, unresponsive to Standard of Care treatment for at least 4 weeks and between ≥ 1 cm2 and ≤ 17.1 cm2 at screening; and between ≥ 1 cm2 and ≤ 12cm2 at the Baseline Visit

Exclusion Criteria:

* Target Ulcer has decreased >30% in size from Screening to Baseline
* Documented history of osteomyelitis at the Target Ulcer location within 6 months preceding the Baseline Visit.
* Patients who are unable to tolerate multi-layer compression therapy.
* Ulcer, which in the opinion of the Investigator is suspicious for cancer.
* Any malignancy within the past 5 years, excluding successfully treated basal cell carcinoma or squamous cell carcinoma without evidence of metastases.
* History of radiation at the Target Ulcer site in previous 12 months prior to Baseline Visit.
* Patients with clinically significant claudication
* Current sepsis
* Patients with known history of significantly compromised immunity for any reason including radiation therapy, chemotherapy or HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Time to complete closure of Target Ulcer | up to 16 weeks
  Time to complete closure of Target Ulcer at any time during the 12-week Treatment Phase. Complete closure is confirmed at two consecutive study visits two weeks apart.

SECONDARY OUTCOMES:
Proportion of complete closure of Target Ulcer | up to 16 weeks
  Proportion of complete closure of Target Ulcer within the Treatment Phase. Complete closure is confirmed at two consecutive study visits two weeks apart.
Percentage change from baseline in Target Ulcer surface area | up to 12 weeks
  Percentage change from baseline in Target Ulcer surface area at the end of the Treatment Phase.
Proportion of Target Ulcer recurrence | up to 24 weeks
  Proportion of Target Ulcer recurrence during the 12-week Follow-Up Phase.

OTHER OUTCOMES:
Adverse Events | up to 24 weeks
  Incidence of adverse events, including overall AEs, AEs related to the CureXcell® and study-ulcer-associated AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kirsner, MD, PhD, Principal Investigator — University of Miami; John Lantis, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center; Robert Snyder, DPM, Principal Investigator — Barry University Clinical Research
Locations (28):
- United States (28):
  - Mesa, Arizona
  - Phoenix, Arizona
  - Carlsbad, California
  - Castro Valley, California
  - Fresno, California
  - Laguna Hills, California
  - Los Angeles, California
  - San Francisco, California
  - Sylmar, California
  - Hialeah, Florida
  - Miami, Florida
  - South Miami, Florida
  - Chicago, Illinois
  - Oak Park, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Las Vegas, Nevada
  - Emerson, New Jersey
  - Summit, New Jersey
  - Toms River, New Jersey
  - New York, New York
  - Chapel Hill, North Carolina
  - Willoughby, Ohio
  - Wyomissing, Pennsylvania
  - Dallas, Texas
  - Lewisville, Texas
  - McAllen, Texas